CLINICAL TRIAL: NCT05145842
Title: The Effect of Combination of Ultrasound and Flouroscopy Guidance in Caudal Epidural Injections on Procedure Time and Radiation Exposure
Brief Title: The Effect of Combination of Ultrasound and Flouroscopy Guidance in Caudal Epidural Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Radiculopathy; Lumbar Disc Herniation; Spinal Stenosis
Keywords: caudal injection; ultrasound; fluoroscopy
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- floroscopy (Active Comparator): 28 patients who have previously been evaluated and planned for caudal epidural injections
  Interventions: Procedure: floroscopy
- ultrasound+fluoroscopy (Experimental): 28 patients who have previously been evaluated and planned for caudal epidural injections
  Interventions: Procedure: ultrasound+fluoroscopy

INTERVENTIONS:
Procedure: floroscopy — After proper antiseptic dressing and draping, sacral hiatus was identified. the position of the needle was confirmed by lateral and anteroposterior fluoroscopic images. The needle was introduced up to S3 level for proper spread of the drug.
  Arms: floroscopy
Procedure: ultrasound+fluoroscopy — After proper antiseptic dressing and draping, the caudal region will be shown in the longitudinal section using sterile probe cover and gel. Under ultrasonographic imaging, the sacrococcygeal ligament will be crossed and the needle will not be advanced any further once the sacral canal is entered. The fluoroscopy phase of the combined imaging will be started and the needle position will be checked by taking an anteroposterior view. The needle tip will be positioned at the sacral 3 level. The needle will be repositioned until the proper position is achieved. The research will be terminated at this point and the time to this stage and the radiation exposure dose will be obtained.
  Arms: ultrasound+fluoroscopy

SUMMARY:
The primary purpose of this study is to asses the effect of caudal epidural injection guided by a combination of ultrasound and fluoroscopy on the duration of the procedure and the amount of radiation exposed during the procedure, compared to the application of only fluoroscopy-guided.

Secondary aims are to reveal the presence of structural variations that prevent injection by examining the morphology of the sacral hiatus by ultrasonography.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. The patients who meet the eligibility requirements will be randomized into two groups in a 1:1 ratio to fluoroscopy and ultrasound+fluoroscopy. Before the procedure, all patients will be scanned with ultrasonography to examine the caudal region morphology.

Processing time will be recorded during injection. "Fluoroscopy time" (sec) and "kerma-area product" (μGy) automatically measured by the fluoroscopy device will be used to evaluate the radiation exposure.

Pre-procedural visual analogue scale (VAS) scores and Oswestry Disability Index (ODI) values were noted all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged> 18 years
* Participation in the study voluntarily
* Diagnosis of radiculopathy caused by spinal stenosis or disc herniation after physical examination and imaging (BT or MRI)

Exclusion Criteria:

* Cauda equina syndrome or rapidly progressing neurological deficit
* previous spine surgery
* local site infection
* history of allergy to local anesthetic and contrast agents
* acute or chronic unstable medical disease
* psychiatric illness
* anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-02-26 (Estimated); Study Completion 2022-05-26 (Estimated)

PRIMARY OUTCOMES:
Processing Time | during the intervention
  The time will be measured by a researcher who will be present in the processing room, using a stopwatch. The chronometer will be started by the researcher with the contact of the needle tip with the skin, in which local anesthetic is used, and the time measurement will be terminated when the spinal treatment needle is withdrawn from the patient.

SECONDARY OUTCOMES:
Fluoroscopy Time | immediately after the intervention
  Fluoroscopy time will be used for the assessment of radiation exposure during the procedure. It is measured automatically by the fluoroscopy device.
Kerma-area Product (μGy) | immediately after the intervention
  Kerma area product is a method of radiation dose monitoring used in radiographic and fluoroscopic studies. It provides an indication of the radiation dose received by a patient. It is measured automatically by the fluoroscopy device.
Visual Analogue Scale | baseline, change from baseline VAS at 2 and 8 weeks after intervention
  Severity of pain was assessed using the standard 10 point VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end
Oswestry Low Back Pain Disability Questionnaire | baseline, change from baseline VAS at 2 and 8 weeks after intervention
  Oswestry Low Back Pain Disability Questionnaire is a scale used to determine the degree of functional disability resulting from low back pain. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Kesikburun, MD, Study Director — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No